CLINICAL TRIAL: NCT06203457
Title: Open-Label Extension Study to Evaluate the Safety of Efgartigimod in Adult Patients With Primary Sjögren's Syndrome (pSS) Who Complete Qualifying Efgartigimod pSS Studies
Brief Title: Open-Label Extension Study to Evaluate the Safety of Efgartigimod in Adult Patients With Primary Sjögren's Syndrome
Acronym: Rho plus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: argenx (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARGX-113-2211
Record Dates: First submitted 2023-11-16; First posted 2024-01-12 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Primary Sjögren's Syndrome
MeSH Terms: interventions — efgartigimod alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- efgartigimod (Experimental): Participants will receive efgartigimod IV infusions
  Interventions: Biological: Efgartigimod

INTERVENTIONS:
Biological: Efgartigimod — Patients receiving efgartigimod infusions

SUMMARY:
Efgartigimod contributes to successfully treat pSS and has the potential to improve disease manifestations by the reduction of IgG autoantibodies in pSS. This open-label extension study will evaluate the long-term safety of efgartigimod in participants with pSS who have completed the treatment period of the qualifying efgartigimod studies (including ARGX-113-2106).

DETAILED DESCRIPTION:
ARGX-113-2211 is a long-term, single-arm, open-label, multicenter extension study of the pSS-qualifying efgartigimod studies designed to evaluate the long-term safety of efgartigimod in adult patients with pSS. Participants will be enrolled from both active and placebo arms of qualifying efgartigimod studies and receive efgartigimod 10 mg/kg over 48 weeks in the extension study without knowledge of their treatment assignment in the qualifying study. Eligible participants must have completed the treatment period of the qualifying study and must not have permanently discontinued the IMP in that study.

ELIGIBILITY:
Inclusion Criteria:

* Is at least the legal age of consent for clinical trials when signing the ICF
* Is capable of providing signed informed consent and complying with protocol requirements
* Agrees to use contraceptive measures consistent with local regulations and the following: WOCBP must have a negative urine pregnancy test at baseline before receiving IMP
* Has completed the qualifying efgartigimod pSS studies and agrees to continue study drug treatment without interruption in the extension study

Exclusion Criteria:

* Clinically significant disease (including newly diagnosed malignancy or cardiovascular disease) or intention to have surgery during the study; or any other medical condition that, in the investigator's opinion, would confound the results of the study or put the participant at undue risk
* Pregnant or intention to become pregnant during the study
* Any severe systemic pSS manifestation that may put the participant at undue risk based on the investigator's opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with (serious) adverse events (of special interest) | up to week 48
Number of participants with with abnormal laboratory test results or vital signs | up to 48 weeks

SECONDARY OUTCOMES:
: Proportion of CRESS (Composite of Relevant Endpoints for Sjögren's Syndrome) responders on ≥ 3 of 5 items at weeks 24 and 48 | up to 48 weeks
  The efficacy of efgartigimod is being assessed based on how the CRESS values change compared to the baseline visits.
Proportion of participants with minimal clinically important improvement from baseline in ESSDAI: improvement of ≥ 3 points in ESSDAI score at weeks 24 and 48 | up to 48 weeks
  ESSDAI is a scoring system/scale - EULAR Sjögren's Syndrome disease activity index (0 to 123). The ESSDAI was designed to measure disease activity in patients with pSS. The lower the scores are, the lower the disease activity is.
Proportion of participants with low disease activity: ESSDAI score of < 5 at weeks 24 and 48 | up to 48 weeks
  ESSDAI is a scoring system/scale - EULAR Sjögren's Syndrome disease activity index (0 to 123). The ESSDAI was designed to measure disease activity in patients with pSS. The lower the scores are, the lower the disease activity is.
Proportion of participants with minimal clinically important improvement from baseline in clinESSDAI: improvement of ≥ 3 points in clinESSDAI score at weeks 24 and 48 | up to 48 weeks
  ClinESSDAI derives from the ESSDAI, and its score provides an accurate evaluation of disease activity independent of B-cell biomarkers. The lower the scores are, the lower the disease activity is.
Proportion of participants with low disease activity: clinESSDAI score of < 5 at weeks 24 and 48 | up to 48 weeks
  ClinESSDAI derives from the ESSDAI, and its score provides an accurate evaluation of disease activity independent of B-cell biomarkers. The lower the scores are, the lower the disease activity is.
Proportion of participants with minimal clinically important improvement from baseline in ESSPRI: decrease of ≥ 1 point or ≥ 15% at weeks 24 and 48 | up to 48 weeks
  ESSPRI is a questionnaire that has been developed to measure self-reported symptoms in participants with pSS. The total global score ranges from 0 to 10, with higher scores indicating more symptoms.
Change from baseline in ESSDAI score at weeks 24 and 48 | up to 48 weeks
  ESSDAI is a scoring system/scale - EULAR Sjögren's Syndrome disease activity index (0 to 123). The ESSDAI was designed to measure disease activity in patients with pSS. The lower the scores are, the lower the disease activity is.
Change from baseline in clinESSDAI score at weeks 24 and 48 | up to 48 weeks
  ClinESSDAI derives from the ESSDAI, and its score provides an accurate evaluation of disease activity independent of B-cell biomarkers. The lower the scores are, the lower the disease activity is.
Change from baseline in ESSPRI score at weeks 24 and 48 | up to 48 weeks
  ESSPRI is a questionnaire that has been developed to measure self-reported symptoms in participants with pSS. The total global score ranges from 0 to 10, with higher scores indicating more symptoms.
Proportion of STAR responders (score of ≥ 5) at weeks 24 and 48 when compared to baseline | up to 48 weeks
  STAR (Sjögren's Tool for Assessing Response) has been developed to assess the efficacy of treatments for pSS.
Percent reduction from baseline in total IgG levels in serum over the 48-week treatment period | up to 48 weeks
Percent reduction from baseline in autoantibodies (Anti-Ro/SS A and Anti-La/SS B) in serum over the 48-week treatment period | up to 48 weeks
Efgartigimod serum concentrations over the 48-week treatment period | up to 48 weeks
Incidence of ADA against efgartigimod over the 48-week treatment period | up to 48 weeks

CONTACTS AND LOCATIONS:
Locations (11):
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Hungary (2):
  - Debreceni Egyetem, Debrecen
  - Vita Verum Medical Egeszsegugyi Szolgaltato Bt., Székesfehérvár
- Poland (8):
  - MCBK SC, Grodzisk Mazowiecki
  - Centrum Medyczne Plejady, Krakow
  - Clinical Research Center Spółka z ograniczoną odpowiedzialnością Medic-R Sp.k., Poznan
  - Centrum Medyczne Pratia Poznan, Skorzewo
  - MICS Centrum Medyczne Warszawa, Warsaw
  - Klinika Reuma Park Sp zoo Sp K, Warsaw
  - Narodowy Instytut Geriatrii, Warsaw
  - FutureMeds sp zoo, Wroclaw

IPD SHARING:
Plan to Share IPD: No